CLINICAL TRIAL: NCT01006005
Title: Adherence-Suppression-Resistance Relationships for Atripla Compared to Historical Antiretroviral Regimens
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: IN-US-177-0106
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections; Adherence
Keywords: HIV; Treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is recruiting 50 patients initiating or switching to Atripla and comparing them to 250 individuals previously followed in a prospective study of HIV+ low income individuals recruited from homeless shelters, single room occupancy hotels and free meal food lines as part of the UCSF Reach Study. Adherence will be measured through monthly unannounced pill counts and electronic medication monitors.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old;
* HIV+;
* Initiating Atripla within 6-months of recruitment;
* Lives in the Tenderloin, South of Market, or Mission District San Francisco;
* Capable of providing informed consent; and
* Willing to complete all study procedures.

Exclusion Criteria:

* Intoxication, cognitive dysfunction or psychosis will preclude potential subjects from informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected, marginally housed
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)